CLINICAL TRIAL: NCT07216547
Title: Post-Operative Trigeminal Pain After Microvascular Decompression for Trigeminal Neuralgia
Status: Not yet recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Gary M. Heir, DMD, Professor, Program and Clinical Director, Rutgers, The State University of New Jersey
Other Study IDs: Pro2025001535
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Trigeminal Neuralgia; Microvascular Decompression Surgery; Post-operative Pain
Keywords: post operative relapse
MeSH Terms: conditions — Trigeminal Neuralgia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the long-term effects of microvascular decompression (MVD) in patients with trigeminal neuralgia (TN). The main question it aims to answer is:

Does undergoing post-operative dental treatment or other orofacial stimulation increase the likelihood of pain relapse after MVD for TN?

Participants who have previously undergone MVD for TN as part of their standard medical care will be asked to complete surveys over phone call. These surveys will focus on their pain experiences, timing, anxiety attacks and nature of any pain relapses, and whether they have received dental treatments or other orofacial interventions during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* MVD post-operative patients with type I Trigeminal Neuralgia.

Exclusion Criteria:

* Atypical (Type II) Facial Pain at presentation, revision surgery.
* Patients who are unable or unwilling to provide informed consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified through a review of the post-operative patient database at Robert Wood Johnson University Hospital in New Brunswick, New Jersey. Eligible subjects are individuals who have undergone initial microvascular decompression (MVD) surgery for trigeminal neuralgia. Medical records will be accessed through the EPIC system, with IRB approval in place
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain control following microvascular decompression (MVD) | Up to 60 months post-surgery
  Pain control will be assessed using the Barrow Neurological Institute (BNI) Pain Scale to evaluate changes in pain severity and relief after MVD.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Heir, DMD, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided